CLINICAL TRIAL: NCT01467323
Title: An Open-labelled, Randomised, Parallel Group, Multicentre, Multinational Efficacy and Safety Comparison of Biphasic Insulin Aspart 30 and Biphasic Human Insulin 30/70 as Meal Related Insulin in a Twice Daily Regimen in Type 1 and Type 2 Diabetic Subjects
Brief Title: Efficacy and Safety of Biphasic Insulin Aspart 30 in Type 1 or Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA/DCD/038
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; biphasic human insulin 30

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: biphasic insulin aspart
- B (Active Comparator)
  Interventions: Drug: biphasic human insulin

INTERVENTIONS:
Drug: biphasic insulin aspart — Injected subcutaneously (under the skin) twice daily
  Arms: A
Drug: biphasic human insulin — Injected subcutaneously (under the skin) twice daily
  Arms: B

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the efficacy and safety of biphasic insulin aspart 30 in subjects with type 1 or type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with insulin requiring type 1 or type 2 diabetes for at least 24 months
* Current treatment with human insulin (either premix of short and long/intermediate acting insulin) in a twice daily treatment regimen preparation and/or self-mix for at least 12 months
* Body mass index (BMI) below or equal to 35.0 kg/m^2
* HbA1c below or equal to 11.0%

Exclusion Criteria:

* Total daily insulin dose at least 1.4 IU/kg
* Treatment with oral hypoglycaemic agents within the month prior to inclusion
* Recurrent severe hypoglycaemia (as judged by the investigator)
* Active proliferative retinopathy
* Impaired renal function with creatinine at least 150 mcmol/l (1.7 mg/dl)
* History of pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 1998-04; Primary Completion 1998-09 (Actual); Study Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin A1c)

SECONDARY OUTCOMES:
8-point blood glucose profiles
Incidence of hypoglycaemic episodes
Occurrence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (35):
- Austria (2):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Vienna
- Germany (15):
  - Novo Nordisk Investigational Site, Anklam
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Cottbus
  - Novo Nordisk Investigational Site, Erkner
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Jena
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Neunkirchen
  - Novo Nordisk Investigational Site, Quakenbrück
  - Novo Nordisk Investigational Site, Rostock
  - Novo Nordisk Investigational Site, Saarlouis
  - Novo Nordisk Investigational Site, Schwedt
  - Novo Nordisk Investigational Site, Ulm
  - Novo Nordisk Investigational Site, Würzburg
- Ireland (2):
  - Novo Nordisk Investigational Site, Cork
  - Novo Nordisk Investigational Site, Dublin
- Novo Nordisk Investigational Site, Bern, Switzerland
- United Kingdom (15):
  - Novo Nordisk Investigational Site, Ayr
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Blackburn
  - Novo Nordisk Investigational Site, Bolton
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Kettering
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Livingstone
  - Novo Nordisk Investigational Site, Newcastle
  - Novo Nordisk Investigational Site, Northampton
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Paisley
  - Novo Nordisk Investigational Site, Watford
  - Novo Nordisk Investigational Site, Whiston

REFERENCES:
- [Result] Boehm BO, Home PD, Behrend C, Kamp NM, Lindholm A. Premixed insulin aspart 30 vs. premixed human insulin 30/70 twice daily: a randomized trial in Type 1 and Type 2 diabetic patients. Diabet Med. 2002 May;19(5):393-9. doi: 10.1046/j.1464-5491.2002.00733.x. PMID 12027927
- [Result] Lindholm A, Jensen LB, Home PD, Raskin P, Boehm BO, Rastam J. Immune responses to insulin aspart and biphasic insulin aspart in people with type 1 and type 2 diabetes. Diabetes Care. 2002 May;25(5):876-82. doi: 10.2337/diacare.25.5.876. PMID 11978684
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com